CLINICAL TRIAL: NCT04708548
Title: Understanding the Long-term Implications of Treatment of Rare Brain Tumours on Health-related Quality of Life: A European Cross-sectional Study
Brief Title: Long Term Implications of Rare Brain Tumours'
Status: Completed | Type: Observational
Sponsor: Galina Velikova (Other)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network); The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor-Investigator, Galina Velikova, Professor., University of Leeds
Organization: University of Leeds (Other)
Other Study IDs: 279885
Record Dates: First submitted 2021-01-07; First posted 2021-01-14 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Quality of Life; Cognitive Impairment; WHO Grade II Oligodendroglial Tumor; WHO Grade III Oligodendroglial Tumor; Long-term Effects of Cancer Treatment; Health-related Quality of Life
MeSH Terms: conditions — Cognitive Dysfunction; Oligodendroglioma | interventions — Quality of Life; Climate Anxiety

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oligodendroglioma (Grade II and III) Patients: Patients diagnosed with a WHO Grade II or III Oligodendroglioma
  Interventions: Other: Health-related Quality of Life; Other: Psychological Distress; Other: Fatigue; Other: Cognitive Functioning

INTERVENTIONS:
Other: Health-related Quality of Life — Health-related quality of life (HRQOL) is an individual's or a group's perceived physical and mental health over time.
Other: Psychological Distress — Measured of the distress experienced by patients
Other: Fatigue — Measure of the extreme tiredness resulting from mental or physical exertion or illness
Other: Cognitive Functioning — Cognitive functioning refers to multiple mental abilities, including learning, thinking, reasoning, remembering, problem solving, decision making, and attention. This will be measured through self-report and cognitive testing.

SUMMARY:
Patients diagnosed with oligodendroglioma with a specific molecular profile represent rare tumour groups (about 10% of adult gliomas) with relatively favourable prognosis (median survival between 8 and 12 years). These patients are often treated with surgery, chemotherapy and/or radiotherapy. However, as patients live for a long period of time, they may also experience long-term toxic side-effects of treatment. The long-term consequences of treatment- and disease-related factors on quality of life and cognitive functioning of these patients are largely unknown. This study aims to investigate quality of life and cognitive functioning in long-term survivors of oligodendroglioma (with IDH mutation and 1p/19q codeletion). This knowledge can support health care professionals prepare patients for any long-term consequences of treatment.

DETAILED DESCRIPTION:
The WHO classification of primary brain tumours has recently been updated and now also takes molecular parameters into account to provide clinicians with more accurate information on the expected disease course and to guide treatment decisions.1 Patients with oligodendrogliomas of WHO grades II or grade III (OII and OIII) defined by IDH mutation and 1p/19q co-deletion represent rare tumour groups (~10% of adult gliomas) with relatively favourable prognosis (median survival 11.9 years for OII and 8.5 years for OIII).2 However, this disease remains life-threatening as over time, all tumours are likely to progress with a more malignant phenotype.

Recent changes in the management of these patients followed after the publication of long-term follow-up data from two landmark studies on OIII carried out by EORTC and RTOG in the 1990s,3, 4 and a RTOG study on low-grade glioma including OII.5 These data suggest that standard treatment should comprise surgical resection of the tumour as feasible followed by radiotherapy and chemotherapy. These studies used radiotherapy doses of 54-60 Gy and PCV (procarbazine, CCNU, vincristine) polychemotherapy. Among high-risk WHO grade II glioma patients, including OII, postoperative temozolomide chemotherapy was not superior in terms of progression-free survival or health-related quality of life (HRQOL) compared to postoperative radiotherapy.6,7 The discussion on whether temozolomide or PCV would be the better chemotherapy in these two patient groups is still ongoing. With patients surviving longer whilst receiving more treatments that may have long-term toxic side-effects, additional questions are raised regarding the effects on HRQOL and cognitive functioning of patients. Indeed, investigating the long-term effects of treatment is listed as a top priority in neuro-oncology research. 8

Preliminary research

The investigational team has almost three decades of research experience in the area of HRQOL and cognitive deficits after glioma treatment. Previous research has found that patients with both low- and high-grade gliomas can experience compromised HRQOL and cognitive functioning, which was generally more pronounced in the high-grade glioma group. However in those with stable, low-grade glioma, HRQOL and cognitive deficits were highly correlated, supporting the notion that even subtle cognitive deficits can affect autonomy in long-term glioma survivors.

While short-term negative effects of chemotherapy on HRQOL are well-documented, longer-term effects of antineoplastic drugs (e.g., bevacizumab) are unknown. Moreover, even low fraction doses of radiotherapy have been shown to have negative consequences for patients' cognitive functioning. WHO grade I and II glioma survivors were assessed on average 12 years after diagnosis and while cognitive functioning had remained stable in patients who had not been treated with radiotherapy, even those who received presumed safe doses (</= 2 Gy) showed a progressive decline in cognitive functioning.9 Moreover, a considerable number of patients showed detectable decline on one or more aspects of HRQOL despite long-term stable disease.6 More recently there have also been investigation into long-term functioning of patients with anaplastic oligo- and oligoastrocytoma. In progression-free patients, HRQOL remained relatively stable whereas cognitive functioning was highly variable across patients, regardless of PCV treatment.7

Despite the recent changes in diagnostics and treatment outlined above, there are no prospective datasets derived from OII/OIII patients treated with the current standards of care. As patients with OII and OIII often receive a range of different treatments for often many years on end, investigating their cognitive functioning and HRQOL becomes ever more important. The long-term consequences of treatment- and disease-related factors on HRQOL and cognitive functioning of patients with OII/OIII 1p/19q codeleted tumours is at present, unknown.

Given the rare occurrence and favourable prognosis of OII/OIII IDH-mutant, 1p/19q codeleted tumours, a cross-European approach is warranted. A collaboration between the EORTC QLG and EORTC BTG provides a unique opportunity to collect pertinent data on how these patients fare after primary treatment. This project aligns with the increased recognition of the issues that cancer survivors face in the long term, both in terms of long-term care needs and in integration in society.

The overall aim of this study is to investigate HRQOL and cognitive functioning of long-term survivors of OII and OIII (with IDH mutation and 1p/19q codeletion). This knowledge can support health care professionals prepare patients for any long-term consequences of treatment, and may even aid in determining to what extent patients might benefit from supportive interventions.

This is a cross-sectional multicentre study, taking place across several European countries. The research co-ordinator and principle investigator are based in Leeds, UK. The co-principle investigator is based in Amsterdam, the Netherlands. Prior to the start of local patient recruitment, each centre will have obtained all relevant ethical and governance approvals.

Patients with OII and OIII with IDH mutation and 1p/19q codeletion diagnosed at least 5 years ago will be recruited, and data on diagnosis and treatment (from medical records), quality of life, mood, fatigue and self-reported cognitive functioning (patient-reported outcomes) and objectively measured cognitive functioning (neuropsychological tests) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed oligodendroglioma WHO grade II or III with IDH mutation and 1p/19q co-deletion
* Diagnosis must have been ≥5 years ago
* Patient is ≥18 years of age
* Willing and able to provide written informed consent

Exclusion Criteria:

* They are expected to be unable to complete consent procedures and/or study outcomes due to legal incompetence or insufficient mastery of the language of the country in which they live as determined by their treating physician.
* They do not provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with a primary brain tumour (histologically confirmed oligodendroglioma) who are patients at participating centres in the United Kingdom, the Netherlands, Germany, France, and other European countries (discussions with countries/centres are ongoing).
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life - EORTC QLQ-C30 | through study completion, an average of 1 year
  To assess the effects of an Oligodendroglioma diagnosis on health related quality of life, The EORTC QLQ-C30 assesses functioning domains (e.g. physical, emotional, role) and common cancer symptoms (e.g. fatigue, pain, nausea/vomiting, appetite loss - the higher the score of each item, the greater the intensity/frequency of the experience e.g., 'Have you had pain?' (1 = not at all, 2 = a little , 3 = quite a bit, 4 = very much)
Disease Specific Quality of Life - EORTC QLQ-BN20 | through study completion, an average of 1 year
  To assess the disease specific quality of life of brain tumour patients. The EORTC QLQ-BN20 consists of 20 items that assess future uncertainty, visual disorder, motor dysfunction, and communication deficit. The higher the score of each item, the greater the intensity/frequency of the experience e.g., 'Did you have difficulty speaking?' (1 = not at all, 2 = a little , 3 = quite a bit, 4 = very much)

SECONDARY OUTCOMES:
Psychological Distress - Hospital Anxiety and Distress Scale (HADS) | through study completion, an average of 1 year
  To measure the psychological distress felt by patients, the HADS is is a 14-item measure designed to assess anxiety and depression symptoms in medical patients, with emphasis on reducing the impact of physical illness on the total score - e.g.- 'I feel tense or 'wound up' (Most of the time, A lot of the time, Time to time, Not at all).
Fatigue - Multidimensional Fatigue Inventory (MFI) | through study completion, an average of 1 year
  To assess the level of fatigue experienced by patients, the Multidimensional Fatigue Inventory (MFI) is a 20-item self-report instrument designed to measure fatigue. - E.G. 'I feel fit' (Yes that is true - No, that is not true (scale going from 1-5, 1 being true, 5 being not true.)
Hopkins Verbal Learning Test - Recall | through study completion, an average of 1 year
  The HVLT-R is a learning test, which consists of 12 words within three semantic groups. The test consists of three acquisition trials in which the administrator reads the words aloud and then asks the participant to repeat as many as they can remember. A delayed recall trial is introduced after 20 min, in which the participant is asked to simply retrieve as many of the words listed in the acquisition trial as he/she can remember. Lower raw scores indicate difficulties with word learning and recall, thus suggesting cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (2):
- Amsterdam UMC, Amsterdam, North Hollan, Netherlands
- Leeds Institute of Medical Research, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boele FW, Frances SM, Darlix A, Ducray F, Cartalat S, Guerdoux E, Tabouret E, Burger MC, Ryden I, Malmstrom A, Vauleon E, Kazda T, Renovanz M, Werner JM, Welsh L, Sanghera P, Dehais C, Desideri I, McBain C, Mehta S, Lord H, Jena R, Foweraker K, Ashkan K, Engelhardt J, Bourg V, Herrlinger U, McLean AL, Hertler C, Haldbo-Classen L, Dahlrot RH, Noel G, Durando X, Hrab I, Razis E, Weller M, Muhic A, Klein M. Health-related quality of life and cognitive functioning in survivors of oligodendroglioma: an international cross-sectional investigation. Neuro Oncol. 2025 Jul 19:noaf172. doi: 10.1093/neuonc/noaf172. Online ahead of print. PMID 40692477
- See also: Research group website/webpage relating to the study — https://pcor.org.uk/understanding-the-long-term-implications-of-treatment-of-rare-brain-tumours-on-health-related-quality-of-life-a-european-cross-sectional-study/